CLINICAL TRIAL: NCT03844087
Title: Effect of Training on the TopSpin360 on Neck Strength and 40-yard Dash Times in Female Varsity Level Athletes
Brief Title: TopSpin360 in Female Varsity Athletes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TopSpin Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 112841
Record Dates: First submitted 2019-02-12; First posted 2019-02-18 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Neuromuscular Strength Training
Keywords: multiplanar, plyometric, neck strength

STUDY DESIGN:
Intervention Model Description: This project will recruit 60 healthy players from Western University's women's soccer and rugby teams. In addition to the team's standard out-of-season baseline testing, participants will have their height, weight, dynamic and static neck strength, neck circumference and 40-yard dash times assessed at baseline. Players will be invited to participate in a 12-week neuromuscular strength training program using the TopSpin360 neuromuscular neck training device. This program will be supervised by a member of the research team 3 days per week in addition to their out-of-season standard training program that does not currently include any exercise specific to the muscles of the neck. Upon completion of the 12 week TopSpin360 training program the study participants will have their weight, neck circumference, dynamic and static neck strength and 40-yard dash times re-assessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- multiplanar neuromuscular training arm (Experimental): The intervention arm will be involved in the training intervention outlined. Briefly, each participant will be asked to train on the TopSpin360 3 times per week for 3-5 sets for the duration of the study. Each set will take roughly 15-30 seconds to perform and training will take part during regularly scheduled training sessions.
  Interventions: Device: Multiplanar neuromuscular training

INTERVENTIONS:
Device: Multiplanar neuromuscular training — See arm description
  Other Names: TopSpin360 training

SUMMARY:
The growing recognition of the short and long-term effects of head-neck trauma on athletes is stimulating the search for preventative measures while improving on-field performance. This study's goal is to evaluate the effect of a 12-week training protocol of the TopSpin360 neuromuscular training device on static and dynamic neck strength and sprinting performance in female varsity level athletes. This study will recruit athletes from the women's varsity soccer and rugby teams. As part of their standard out of season testing, they will have their static and dynamic neck strength, neck girth and 40 yard dash times assessed at inception into the study. The athletes will then be invited to participate in the TopSpin360 training program. This program incorporates training sessions on the TopSpin360 of 3-5 sets of 50 revolutions in each direction of clockwise and counterclockwise three times a week to improve static and dynamic neck strength but not sprint performance specifically. The sessions last 10-15 minutes and will run for 12 weeks. Members of the research team will supervise these training sessions 3 days per week as an addition to their out of season training program. Neck girth, static and dynamic neck strength and 40 yard dash times will be reassessed after the 12 week training intervention. The study hypothesis is that training on the TopSpin360 will result in improved static and dynamic neck strength and improved 40-yard dash times. A secondary hypothesis is that the change in neck strength will be positively associated with the change in 40-yard dash times, aligning with an emerging theory of athletic performance related to dynamic control of the entire kinetic chain including the neck. Routine re-evaluation of neck strength throughout the duration of the 12-week program will provide additional information on the trajectory of training effects and estimates of time-to-peak performance.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the effect of training using a new neck protocol on two primary outcomes: neck strength (both dynamic and static) and 40-yard dash times in a group of healthy university-aged female athletes.

The secondary purposes are to 1. explore the temporal components of performance increase, notably the trajectory of training effects. 2. explore the carryover effects of training between performance metrics by evaluating the associations between dynamic performance on the training device, isometric neck strength and 40-yard dash times. 3. examine the effects of the training program on neck girth. 4. As a sub-purpose for further research, capture available data to explore a potential relationship between previous concussion history and static and dynamic neck strength during training.

All participants will be informed of the study through an email from the team's coaching staff prior to their team's out of season baseline testing at the Kirkley Training Centre at TD (Toronto Dominion) Stadium and Thompson Arena indoor track. Interested athletes will be given an email address of one of the research team to contact for further information. Those who consent will undergo a screening protocol to identify any gross cervical dysfunction prior to a baseline evaluation that includes static and dynamic neck strength assessment, neck girth measurement and 40 yard dash time. A member of the research team (physiotherapy student) will perform the screening protocol. This involves assessing full active range of motion in 6 planes of movement, no pain during the 4 quadrants 'combined planes' test, no pain with the Spurling's cervical compression test (Tong, Haig, & Yamakawa, 2002). Static neck strength will be assessed by a neck strength assessment protocol as described by Versteegh et. al. (Versteegh, Beaudet, Greenbaum, Hellyer, Tritton, Walton, 2015). Briefly, this involves having the participant hold a handheld dynamometer (force measuring device) with a soft foam contact area that is placed against the head at different points (front, back, and each side one at a time). The participant applies their own resistance with their arm(s) as they push maximally into the dynamometer with encouragement from the researchers. Peak force is held in each direction for 3 seconds and peak strength values are recorded in each direction (8 total tests). These 8 test values will be summed and divided by 8 to provide a composite neck strength score as the primary outcome measure and dependent variable for data analysis.

Following baseline testing, each participant will be familiarized with the TopSpin360. The TopSpin360 is a neuromuscular training device that is akin to a 'hula hoop' for the neck, the protocol leverages self-generated centripetal force created by using the neck to keep a weighted arm rotating about the top of a custom-fitted helmet. Each participant will have the properly sized device securely fastened to their head using the provided chin straps. They will then familiarize themselves with the exercise motion of getting the small weight to spin about the centrally mounted axis in both directions. Because the weight is relatively light, the resistance to the muscles is only produced by the centripetal force created by the spinning weight. Once they are comfortable with the exercise patterning they will perform 50 timed revolutions in each direction of clockwise and counter-clockwise. These evaluation sets will be timed (metric 1) and the peak velocity achieved for each set (metric 2) will be recorded. Neck girth will be measured using a flexible measuring tape at the level of the thyroid cartilage. Participants will have their height measured using a measuring tape against a wall, weight will be measured using the standard scale at the Kirkley Centre and participants will be asked about their previous concussion history.

After baseline neck strength assessments are performed, the participants will proceed to Thompson arena. After performing an appropriate warm-up administered by the strength and conditioning coach, the participants will complete a 40-yard dash at the indoor track. This sprint will be timed using the Western varsity athlete's electronic sprint timing system. All data will be entered into a Microsoft Excel worksheet using a unique subject number. The single master list linking the subject's name and unique number will be stored separately from the de-identified data file. Participants will also be asked if they have ever had a previous concussion and if so, how many have they had and if they have had any in the past 12 months.

The participant will then be scheduled to attend an initial training session with one of the student researchers. This initial training session will go through the neuromuscular training program (roughly 20-30 minutes for familiarization with the program). After this session, the participants and the student researchers will create a training schedule for the study program with an effort to accommodate each participant's out of season training schedule. The program will be three training sessions per week for 12 weeks, performed in conjunction with their current out of season training program. Each of these additional training sessions will last 10-15 minutes.

The neuromuscular training program is broken up into four different phases: Foundation, Stability, Balance, and Movement. Each phase progresses the TopSpin360 exercises over 3 week periods from seated, to standing, to single leg, and lastly squats and lunges. Each training session will involve performing 3 to 5 sets of 50 revolutions in each direction of clockwise and counter-clockwise as described above. The participants will be encouraged to perform each set as quickly as they are able (on average 20-45 seconds per set). Between each set the participants will be allowed to rest for 1-2 minutes. During these training sessions, the peak velocity achieved for each direction and the time to complete each set will be recorded. This protocol will be continued for the remaining sessions until program completion after the 36th session or the end of 12-weeks, whichever comes first. Upon completion of the 12-week training session, participants will be re-evaluated using the same assessment as the baseline protocol described above. This includes the time required to perform 50 revolutions clockwise and counter-clockwise, peak velocity achieved on the device along with re-evaluating their isometric neck strength, neck circumference and body weight. Re-assessment of the 40 yard dash will be completed at Thompson arena as it was at baseline. During the course of the study, all participants will be encouraged to participate in their regular physical activity.

This study is largely exploratory in nature, meaning sample sizes are being estimated erring on the side of conservativeness and feasibility. Our prior pilot study revealed a moderate effect size on isometric neck strength (Hedge's d = 0.68) in a sample of male varsity football players over a 7-week training period, though we cannot assume this same effect will translate to a sample of female varsity soccer and rugby players, hence part of the motivation for this study. We anticipate the analysis requiring the largest sample will be the association between change in neck strength and change in sprint performance. There are some potential sources of noise here including the test-retest reliability of the sprint performance that we need to consider. We are also unsure on the variance expected in the change in sprint performance which will influence the magnitude of correlation between it and change in neck performance. If we estimate a small-to-medium association between the two change scores of r = 0.40 (coefficient of determination = 0.16), desiring a correlation of 80% power and accepting a 5% two-tailed alpha error rate, then g*power software indicates a sample size of n = 46 participants, however this does not include some of the unknown variables. As there are 60 athletes across the two (soccer and rugby) teams we will aim to recruit all 60, a strategy that will also mean we do not preclude any player from participating in what we suspect will be a beneficial intervention.

The primary hypothesis: Participation in the training protocol will improve static and dynamic neck strength and 40 yard dash times. Analysis will occur through a repeated measures ANOVA where time is the independent variable and neck strength (static and dynamic) and 40-yard dash time are the dependent variables. Significant main effects will be explored using Tukey's post-hoc to identify significant interactions between the three dependent variables.

It is also anticipated that higher adherence to the training program may be associated with greater improvements in neck strength and 40 yard sprint performance. Linear regression will be used to analyze if higher adherence is associated with greater improvements in the dependent variables.

Secondary hypothesis 1: To explore the temporal components of performance increases. This will be analyzed graphically by plotting the peak RPM (revolution per minute) achieved in each training session with time.

Secondary hypothesis 2: There will be a strong association between static and dynamic neck strength after the training period. This will be analyzed through Pearson's r correlation coefficient between the peak RPM achieved and the composite neck strength score post training.

Secondary hypothesis 3: Greater adherence to the training program will lead to greater improvements in neck girth. This will be analyzed through paired t-tests of neck girth values pre training to post training and through linear regression between changes in neck girth and training program adherence.

Secondary hypothesis 4: The participants with a prior history of concussion will have lower static and dynamic neck strength than players with no history of concussion. Analysis will occur through independent t-test of composite static neck strength between players with a history of concussion and players with no history of concussion. Likewise for dynamic neck strength values.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults on Western University's women's soccer and rugby teams

Exclusion Criteria:

* those who are not medically cleared to participate in out of season training, or anyone under the age of 18

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in static neck strength as measured using a handheld dynamometer | Change from Baseline Static Neck Strength after 12 weeks of training
  Multiplanar static neck strength
Change in Dynamic neck strength | Change from Baseline Performance in Dynamic Neck Strength after12 weeks of training
  Performance on the TopSpin360
Change in 40 yard dash time | Change from Baseline 40 yard dash time after 12 weeks of training
  time to sprint 40 yards

SECONDARY OUTCOMES:
Change in Neck girth | Change in Neck Girth after 12 weeks of training
  neck girth measurement
Relationship between self-declared concussion history and static and neck strength | As measured at Baseline
  Independent t-tests between average static and dynamic neck strength of those with a history of concussion compared to the average static and dynamic neck strength of those without a history of concussion

CONTACTS AND LOCATIONS:
Overall Officials: David M Walton, PhD, Principal Investigator — Western University
Locations (1):
- Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Versteegh T, Beaudet D, Greenbaum M, Hellyer L, Tritton A, Walton D. Evaluating the reliability of a novel neck-strength assessment protocol for healthy adults using self-generated resistance with a hand-held dynamometer. Physiother Can. 2015 Winter;67(1):58-64. doi: 10.3138/ptc.2013-66. PMID 25931654
- [Background] Tong HC, Haig AJ, Yamakawa K. The Spurling test and cervical radiculopathy. Spine (Phila Pa 1976). 2002 Jan 15;27(2):156-9. doi: 10.1097/00007632-200201150-00007. PMID 11805661